CLINICAL TRIAL: NCT06440135
Title: An Open Label Phase I Study of Ziftomenib as Maintenance Therapy Following Allogeneic Hematopoietic Cell Transplantation
Brief Title: Ziftomenib Maintenance Post Allo-HCT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Zachariah Michael DeFilipp, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-096
Record Dates: First submitted 2024-03-05; First posted 2024-06-03 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia in Remission; NPM1 Mutation; KMT2A Rearrangement
Keywords: Acute Myeloid Leukemia; Allogeneic hematopoietic cell transplantation (HCT); Allo-HCT; NPM1 Mutation; KMT2A Rearrangement
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ziftomenib (Experimental): Participants will begin treatment 30 to 90 days after allo-HCT and only after disease remission is confirmed, and treatment will continue for up to 12 months. All participants will receive ziftomenib. Participants will undergo allo-HCT as a part of their standard care.
  Participants will undergo the following procedures:
  * Screening
  * Allo-HCT (standard care), including pre and post-treatment as a part of standard care
  * 30 - 90 days after allo-HCT, participants will take the study drug orally once per day for up to 12 28-day cycles
  * End of treatment visit
  * Follow-up data will be collected every 3 months for 24 months from the start of treatment
  Interventions: Drug: Ziftomenib

INTERVENTIONS:
Drug: Ziftomenib — Taken orally once per day
  Other Names: KO-539

SUMMARY:
The purpose of this study is to test the safety, effects, and recommended dose of an investigational drug, ziftomenib, in addition to the standard treatment on blood cancer with Allogeneic Hematopoietic Cell Transplantation (allo-HCT). This study plans to learn more about ziftomenib, which targets and inhibits negative interactions within cancer cells related to AML, when given after allo-HCT, to determine if it improves outcomes following allo-HCT.

The name of the study drug involved in this study is:

• Ziftomenib

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, phase I study of ziftomenib as maintenance therapy following allogeneic hematopoietic cell transplantation (HCT). This study is testing whether ziftomenib, combined with the standard allo-HCT treatment, is safe and effective in treating blood cancer. This study will test if ziftomenib improves outcomes after allo-HCT.

The study drug is given after the allo-HCT, in combination with standard treatment and aftercare.

This study consists of 2 parts:

Part A (Dose Escalation): The investigators are looking to find the highest dose of the study intervention that can be administered safely without severe or unmanageable side effects, not everyone who participates in this research study will receive the same dose of the study intervention. The dose given will depend on the number of participants who have been enrolled prior and how well the dose was tolerated. Once determined, this highest dose will then be used in the dose expansion part of the study.

Part B (Expansion Cohort): Participants will be treated at the respective dose as determined during Part A(Dose Escalation).

Ziftomenib administered after allo-HCT may work to enhance graft-versus-leukemia effects, selectively target residual leukemic cells, or suppress leukemic stem cells, among other mechanisms. The U.S. Food and DrugAdministration (FDA) has not currently approved ziftomenib as a treatment for any disease but it is being studied in Phase 1/2 interventional clinical trials for participants with relapsed or refractory acute myelogenous leukemia.

The estimated length of the study is 2 years. Participants will begin treatment 30 to 90 days after allo-HCT, and treatment will continue for up to 12 months. Then they will be followed for 12 to 24 months after study treatment ends.

It is expected that about 22 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Pathologically confirmed diagnosis of acute myeloid leukemia (AML).
* Complete remission (CR) or complete remission with incomplete count recovery (CRi) at screening.

  * Complete remission (CR):

    * no circulating blasts in peripheral blood and <5% blasts in bone marrow
    * no extramedullary disease
    * platelet count ≥100 x 10(9)/L and/or absolute neutrophil count ≥1000/µL
  * Complete remission with incomplete count recovery (CRi):

    * no circulating blasts in peripheral blood and <5% blasts in bone marrow
    * no extramedullary disease
    * platelet count <100 x 10(9)/L and/or absolute neutrophil count <1000/µL
* Presence of at least one of the following molecular mutations:

  * KMT2A rearrangement

    * Eligibility and enrollment will be based on local mutational testing.
    * The presence of a KMT2A rearrangement (excluding partial tandem duplication [PTD]) at the time of initial diagnosis or any other time thereafter is sufficient.
    * Participants may receive additional treatment for AML between consent and transplant.
  * NPM1 mutation

    * Eligibility and enrollment will be based on local mutational testing.
    * For participants being transplanted in CR1, the presence of a NPM1 mutation at screening is necessary for the purposes of eligibility.
    * For participants being transplanted in greater than or equal to CR2, the presence of a NPM1 mutation at the time of consent is not necessary for eligibility and its presence at the time of initial diagnosis or any other time thereafter is sufficient.
    * Participants may receive additional treatment for AML between consent and transplant.
* Treatment with a menin inhibitor prior to transplant is permitted. However, patients who experienced AML relapse or progression while being treated with a menin inhibitor prior to transplant are ineligible.
* Will undergo first allogeneic HCT for their malignancy.
* Transplantation will be performed with the use of conventional myeloablative (MAC) or reduced intensity conditioning (RIC).
* HCT Donor will be one of the following:

  * 5/6 or 6/6 (HLA-A, B, DR) matched related donor
  * 7/8 or 8/8 (HLA-A, B, DR, C) matched unrelated donor. Matching in the unrelated setting must be at the allele level.
  * Haploidentical related donor, defined as ≥ 3/6 (HLA-A, B, DR) matched
  * ≥ 4/6 (HLA-A, B, DR) umbilical cord blood (UCB). Matching in the UCB setting is at the antigen level. Recipients may receive either one or two UCB units. In the case of 2 UCB units, both units must have been at least 4/6 matched with the recipient.
* Any non-investigational GVHD prophylaxis regimen is allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Participants must have normal organ and function as defined below:

  * AST (SGOT), ALT (SGPT) and Alkaline phosphatase < 3x institutional upper limit of normal (ULN)
  * Total bilirubin < 1.5 x institutional ULN (with the exception of subjects with a history of Gilbert's syndrome, for which the total bilirubin must be < 5 x ULN)
  * Calculated creatinine clearance ≥ 30 mL/min (Cockcroft-Gault formula)
* LVEF must be ≥50%, as measured by MUGA scan or echocardiogram.
* Female patients of childbearing potential must have a negative pregnancy test, as measured by serum or urine testing.
* The effects of ziftomenib on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) during the entire study treatment period and through 6 months after the last dose of treatment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of other malignancy(ies) unless

  * the participant has been disease-free for at least 2 years and is deemed by the investigator to be at low risk of recurrence of that malignancy, or
  * the cancer has been deemed indolent with no progression over the last 2 years, and deemed by the investigator to be at low risk for further progression during the course of study and follow-up
  * the only prior malignancy was cervical cancer in situ and/or basal cell or squamous cell carcinoma of the skin
* Known diagnosis of active hepatitis B or hepatitis C
* Current or history of congestive heart failure New York Heart Association (NHYA) class 3 or 4, or any history of documented diastolic or systolic dysfunction (LVEF < 50%, as measured by multigated acquisition (MUGA) scan or echocardiogram)
* Current or history of ventricular or life-threatening arrhythmias or diagnosis of long-QT syndrome
* Systemic uncontrolled infection
* Known dysphagia, short-gut syndrome, gastroparesis, or other condition(s) that limits the ingestion or gastrointestinal absorption of drugs administered orally
* Uncontrolled hypertension (systolic blood pressure [BP] > 180 mmHg or diastolic BP > 100 mmHg)
* QTc interval (i.e., Friderica's correction [QTcF]) ≥ 480 ms or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) at screening
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* Persons who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (Dose Escalation) | 28 days
  Defined as the highest dose level at which 1 or 0 of 6 patients experience a Dose Limiting Toxicity (DLT). Toxicities will be graded and documented according to NCI CTCAE version 5.0.
  A non-hematologic DLT is any grade 3 adverse event (AE) lasting >72 hours or any grade greater than or equal to 4 AE that is at least possibly related to the study drug with exceptions.
  Any ≥ grade 2 non-hematologic toxicity that the participant finds intolerable or renders the participant unable to take 75% or more of the assigned doses (e.g. multiple dose interruptions) during the first cycle will be considered a DLT.

SECONDARY OUTCOMES:
Occurrence of ziftomenib-related toxicities | Day 0 to last treatment dose, up to 336 days
  Defined as ziftomenib-related toxicities detected and categorized according to severity. Toxicities will be graded and documented according to NCI CTCAE version 5.0.
Incidence of acute Graft versus Host Disease (GVHD) during treatment | Day 0 to end of treatment visit, up to 366 days (336 days of treatment + 30 days end of treatment)
  Defined as cumulative incidence of acute GVHD from start of ziftomenib in subjects receiving maintenance therapy after allogeneic HCT. Clinical stage and grade of acute graft-versus-host-disease (GVHD) is based on MAGIC Criteria (Harris 2016). The incidence of acute GVHD grade II-IV and grade III-IV will be estimated for each treatment group using the cumulative incidence estimate, treating death prior to acute GVHD as a competing event.
Incidence of chronic Graft versus Host Disease (GVHD) during treatment | Day 0 to end of treatment visit, up to 366 days (336 days of treatment + 30 days end of treatment)
  The incidence of chronic GVHD will be estimated for each treatment group using the cumulative incidence estimate, treating death prior to chronic GVHD as a competing event. Chronic GVHD will be assessed as per the 2014 National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease (Jagasia 2015).
Non-relapse mortality (NRM) | Day 0 to end of treatment visit, up to 1086 days (336 days of treatment + 30 days end of treatment + 24 months follow-up))
  The incidence of non-relapse mortality will be estimated for each treatment group using the cumulative incidence estimate, treating disease relapse or progression as a competing event. AML treatment response is based on 2022 ELN recommendations (Dohner 2022).
Leukemia-Free Survival (LFS) | Day 0 to end of treatment visit, up to 1086 days (336 days of treatment + 30 days end of treatment + 24 months follow-up))
  Leukemia-Free Survival is defined as the time from first dose of study drug to the earlier of leukemia relapse or death due to any cause. Participants alive and leukemia-free are censored at the date of last disease evaluation. AML treatment response is based on 2022 ELN recommendations (Dohner 2022).
Overall Survival (OS) | Day 0 to end of treatment visit, up to 1086 days (336 days of treatment + 30 days end of treatment + 24 months follow-up))
  Overall Survival is defined as the time from first dose of study drug to the date of death due to any cause. Participants who are alive at the analysis / cutoff date will be censored at the last contact date.
GVHD-free, relapse-free survival (GRFS) | Day 0 to end of treatment visit, up to 1086 days (336 days of treatment + 30 days end of treatment + 24 months follow-up))
  GVHD, relapse-free survival is defined as the time from first dose of study drug to the earlier of grade III-IV acute GVHD, chronic GVHD requiring systemic immune suppression, leukemia relapse or death due to any cause. Participants alive and without one of these three events are censored at the date of last disease evaluation. AML treatment response is based on 2022 ELN recommendations (Dohner 2022).
Proportion of successfully screened that do not reach study treatment | 30 days (Screening to Day 0)
  Defined as proportion of subjects who successfully screen for study prior to transplantation but who do not reach the maintenance phase due to transplant-related morbidity or mortality.
Plasma Concentration of ziftomenib and metabolites | Up to 62 days (Cycle 1 Day 1 - Cycle 3 Day 1 (+/- 5 days)
  Characterize the pharmacokinetics (PK) of ziftomenib and metabolites when ziftomenib is given as maintenance therapy after allogeneic HCT by measuring the plasma concentration of ziftomenib and metabolites.
Plasma Concentration of oral immunosuppressive agents and ziftomenib | Up to 34 days (Day -7 to -14 after HCT prior to co-administration and on Cycle 1 Day 1 and Day 15 (+/- 5 days) of co-administration)
  Assess PK drug-drug interaction between ziftomenib and oral systemic immunosuppressive agents performed by measuring plasma concentrations.
Number of Participants with Treatment-Related Adverse Events | Day 0 to end of treatment visit, up to 366 days (336 days of treatment + 30 days end of treatment)
  The severity/intensity of adverse events will be graded based upon the subject's symptoms according to the current active minor version of the Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0). All participants will be followed and assessed for adverse events 30 days after removal from protocol therapy or until death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Zachariah DeFilipp, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Zachariah DeFilipp, MD. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation